CLINICAL TRIAL: NCT01370421
Title: Prediction of Outcomes Following Total Knee Replacement
Acronym: POKR
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert Edwards, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2010p000978
Record Dates: First submitted 2011-06-02; First posted 2011-06-10 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee OA patients undergoing Total Knee Arthroplasty (TKA): Participants will be 45 years or older, diagnosed with Osteoarthritis of the knee and be scheduled for a unilateral total knee replacement surgery.

SUMMARY:
This is an observational study (not a treatment study) of pain and physical functioning after total knee replacement. The study includes 5 visits, 1 before surgery and 4 after surgery. You may be eligible if you are 50 or older,will soon be undergoing knee replacement surgery, do not have a serious heart condition or certain other medical conditions, and are not taking certain types of medications. The study includes evaluation of peoples' pain, physical functioning, medication use, and physiological responses to sensory stimuli such as heat and cold.

DETAILED DESCRIPTION:
This is an observational study (not a treatment study) of pain and physical functioning after total knee replacement. The study includes 5 visits, 1 before surgery and 4 after surgery. The last visit will be about 1 year after surgery. You may be eligible if you are 50 or older, will soon be undergoing knee replacement surgery, do not have a serious heart condition or certain other medical conditions, and are not taking certain types of medications. The study includes evaluation of peoples' pain, physical functioning, medication use, and physiological responses to sensory stimuli such as heat and cold.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Meet the American College of Rheumatology criteria for knee osteoarthritis
* Scheduled to undergo total knee arthroplasty
* Facility with the English language that is adequate to complete study procedures

Exclusion Criteria:

* Cognitive impairment preventing completion of study assessment procedures
* Myocardial infarction within the past 12 months
* Severe raynaud's or severe neuropathy
* Active vasculitis or severe peripheral vascular disease
* Current infection
* Use of oral steroids
* Recent history of substance abuse or dependence
* Confirmed diagnosis of periodic limb movement disorder or restless legs syndrome
* Systemic inflammatory or autoimmune disorders such as rheumatoid arthritis, lupus, etc.
* Known anemia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants for this study will be recruited via flyers posted in hospital clinics, on electronic announcement boards and various other media mediums. Potential subjects will be informed about the study purpose and procedures when they call, and interested subjects will then go through a telephone screening.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | 6 months
  A widely-used measure of pain severity and pain interference. Pain severity and pain interference scores range from 0-10 (0= no pain / no pain interference and 10= severe pain / pain interference).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months
  A widely-used, OA-specific measure of pain, function, and stiffness. WOMAC Pain scores range from 0-50, with 0= no pain and 50= severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States